CLINICAL TRIAL: NCT03347188
Title: A Phase 2, Multicenter, Randomized, Proof-of-Concept, Double-Blind, Placebo-Controlled, Parallel-Group Study, Including an Open-Label Period, Evaluating the Efficacy and Safety of 1 Subcutaneous Dose Regimen of Fremanezumab for the Treatment of Posttraumatic Headache (PTH)
Brief Title: A Study to Test if Fremanezumab Reduces Headache in Participants With Posttraumatic Headache (PTH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TV48125-CNS-20024
Expanded Access: NCT03539393 (Available)
Record Dates: First submitted 2017-11-14; First posted 2017-11-20 (Actual); Results first posted 2021-03-26 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Post-Traumatic Headache
Keywords: posttraumatic headache (PTH)
MeSH Terms: conditions — Post-Traumatic Headache | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fremanezumab (Experimental): Participants will receive fremanezumab 675 milligrams (mg) administered as 3 subcutaneous (SC) injections (225 mg/1.5 milliliters [mL] each) at randomization (Week 0), Weeks 4, and 8 during the DB treatment period. Participants who complete the DB treatment period and continue into the OL treatment period will receive fremanezumab 675 mg administered as 3 SC injections (225 mg/1.5 mL each) at Weeks 12, 16, and 20 during the OL treatment period.
  Interventions: Drug: Fremanezumab
- Placebo (Placebo Comparator): Participants will receive placebo matching to fremanezumab administered as 3 SC injections (1.5 mL each) at randomization (Week 0), Weeks 4, and 8 during the DB treatment period. Participants who complete the DB treatment period and continue into the OL treatment period will receive fremanezumab 675 mg administered as 3 SC injections (225 mg/1.5 mL each) at Weeks 12, 16, and 20 during the OL treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fremanezumab — Fremanezumab will be administered per dose and schedule specified in the arm.
  Other Names: TEV-48125
  Arms: Fremanezumab
Drug: Placebo — Placebo matching to fremanezumab will be administered per schedule specified in the arm.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the safety and efficacy of fremanezumab in adult participants aged 18 to 70 years, inclusive, for the prevention of PTH. The study will include a double-blind (DB) treatment period (12 weeks) and an open-label (OL) treatment period (12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* The participant has a body weight greater than or equal to (≥) 45 kilograms (kg).
* Traumatic injury to the head has occurred, defined as a structural or functional injury resulting from the action of external forces.
* The participant has a diagnosis of PTH.
* The participant is not using preventive medications for headache.
* Women of childbearing potential whose male partners are potentially fertile (that is, no vasectomy) must use highly effective birth control methods for the duration of the study and for 30 weeks after the last study drug administration. Men must be sterile or, if they are potentially fertile or reproductively competent (that is, not surgically or congenitally sterile) and their female partners are of childbearing potential, must use, together with their female partners, acceptable birth control methods for the duration of the study and for 30 weeks after the last study drug administration.

NOTE- Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* The participant has a previous history of brain imaging showing evidence of intracerebral hemorrhage, subdural or epidural hematomas, or subarachnoid hemorrhage as a consequence of the traumatic head injury. Brain images with structurally insignificant changes, as discussed and approved by the sponsor, will be reviewed by the sponsor on a case-by-case basis.
* The participant has PTH attributed to craniotomy.
* The participant has whiplash and subsequent headache but no history of head injury or concussion.
* The participant is using analgesic medications containing opioids (including codeine) or a barbiturate on average more than 15 days per month.
* The participant has had exposure to a monoclonal antibody (mAb) targeting the calcitonin gene-related peptide (CGRP) pathway (erenumab, eptinezumab, galcanezumab, and fremanezumab) during the 6 months prior to the day of the screening visit.
* The participant is currently being treated with onabotulinumtoxinA (for example, Botox, Dysport, Xeomin) application in the head or neck or received any such injection during the 3 months prior to the screening visit.
* The participant has been implanted with any electronic devices for headache prevention during the 3 months prior to the screening visit or is currently using any implanted or externally applied stimulator or device.
* The participant has been treated with a nerve block for head and/or neck during the 3 months prior to the screening visit.
* The participant is a pregnant or lactating woman or plans to become pregnant during the study.

NOTE- Additional criteria apply, please contact the investigator for more information.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (33):
- United States (33):
  - Teva Investigational Site 14065, Phoenix, Arizona
  - Teva Investigational Site 14069, Scottsdale, Arizona
  - Teva Investigational Site 14048, Little Rock, Arkansas
  - Teva Investigational Site 30236, Little Rock, Arkansas
  - Teva Investigational Site 14052, Long Beach, California
  - Teva Investigational Site 14053, Los Angeles, California
  - Teva Investigational Site 14060, San Diego, California
  - Teva Investigational Site 14054, San Francisco, California
  - Teva Investigational Site 14045, Fairfield, Connecticut
  - Teva Investigational Site 14063, Miami, Florida
  - Teva Investigational Site 14041, North Miami, Florida
  - Teva Investigational Site 14056, Tampa, Florida
  - Teva Investigational Site 14057, Riverwoods, Illinois
  - Teva Investigational Site 14067, Indianapolis, Indiana
  - Teva Investigational Site 14058, Louisville, Kentucky
  - Teva Investigational Site 14061, Waltham, Massachusetts
  - Teva Investigational Site 14051, Kansas City, Missouri
  - Teva Investigational Site 14043, Springfield, Missouri
  - Teva Investigational Site 14046, St Louis, Missouri
  - Teva Investigational Site 14119, Albany, New York
  - Teva Investigational Site 14229, Amherst, New York
  - Teva Investigational Site 14047, New York, New York
  - Teva Investigational Site 14118, The Bronx, New York
  - Teva Investigational Site 14114, Durham, North Carolina
  - Teva Investigational Site 14059, Salisbury, North Carolina
  - Teva Investigational Site 14049, Portland, Oregon
  - Teva Investigational Site 14064, Philadelphia, Pennsylvania
  - Teva Investigational Site 14040, Pittsburgh, Pennsylvania
  - Teva Investigational Site 14230, Nashville, Tennessee
  - Teva Investigational Site 14055, Dallas, Texas
  - Teva Investigational Site 14050, Waco, Texas
  - Teva Investigational Site 14113, Spokane, Washington
  - Teva Investigational Site 14044, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Fremanezumab: Participants received fremanezumab 675 milligrams (mg) administered as 3 subcutaneous (SC) injections (225 mg/1.5 milliliters [mL] each) at randomization (Week 0), Weeks 4, and 8 during the double-blind (DB) treatment period. Participants who completed the DB treatment period and continued into the open-label (OL) treatment period received fremanezumab 675 mg administered as 3 SC injections (225 mg/1.5 mL each) at Weeks 12, 16, and 20 during the OL treatment period.
- Placebo: Participants received placebo matched to fremanezumab administered as 3 SC injections (1.5 mL each) at randomization (Week 0), Weeks 4, and 8 during the DB treatment period. Participants who completed the DB treatment period and continued into the OL treatment period received fremanezumab 675 mg administered as 3 SC injections (225 mg/1.5 mL each) at Weeks 12, 16, and 20 during the OL treatment period.
Period: Double-blind (DB) Period (12 Weeks)
Arm/Group | Fremanezumab | Placebo
Started | 44 | 43
Received at Least 1 Dose of Study Drug | 43 | 43
Full Analysis Set (FAS) (Received at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment on primary endpoint.) | 42 | 43
Completed | 29 | 26
Not Completed | 15 | 17
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 4 | 8
Not completed — Lost to Follow-up | 7 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Other than specified | 1 | 2
Period: Open-label (OL) Period (12 Weeks)
Arm/Group | Fremanezumab | Placebo
Started | 35 | 35
Entered in OL Period for Anti-drug Antibody (ADA) Only | 26 | 28
Received at Least 1 Dose of Study Drug | 9 | 7
Completed | 8 | 6
Not Completed | 27 | 29
Not completed — Entered for ADA assessment only, not treated | 26 | 28
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other than specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Fremanezumab: Participants received fremanezumab 675 mg administered as 3 SC injections (225 mg/1.5 mL each) at randomization (Week 0), Weeks 4, and 8 during the DB treatment period. Participants who completed the DB treatment period and continued into the OL treatment period received fremanezumab 675 mg administered as 3 SC injections (225 mg/1.5 mL each) at Weeks 12, 16, and 20 during the OL treatment period.
- Total: Total of all reporting groups
Arm/Group | Fremanezumab | Placebo | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (13.01) | 43.8 (14.48) | 43.2 (13.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 19 | 18 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 40 | 38 | 78
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 41 | 39 | 80
  Race: Black or African American | 3 | 1 | 4
  Race: Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  Race: Other | 0 | 2 | 2
Number of Headache Days of at Least Moderate Severity [Mean (Standard Deviation); unit: days] — Population: 'Number analyzed' signifies participants evaluable for this baseline measure.
  days
    number analyzed (Participants) | 43 | 43 | 86
    (all) | 18.7 (7.03) | 18.5 (6.12) | 18.6 (6.56)

OUTCOME MEASURES:

1. Primary Outcome: DB Period: Mean Change From Baseline in Monthly Average Number of Headache Days of at Least Moderate Severity During the 12-Week Treatment Period After the First Dose of Fremanezumab
Description: A headache day was defined as a day when a participant reported a headache of at least moderate severity. Monthly averages were derived and normalized to 28 days equivalent by the following formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in the e-diary over the relevant period) * 28. The change was calculated as post-baseline value - baseline value. Least square (LS) mean was calculated using analysis of covariance (ANCOVA) model with the duration of post traumatic headache history (less than 12 month since the brain injury or greater or equal to 12 month since the brain injury) and treatment as fixed effects and the baseline monthly average number of headache days of at least moderate severity as a covariate.
Time Frame: Baseline (Day -28 to Day -1), up to Week 12
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of the study drug and had at least 1 post-baseline efficacy assessment on the primary endpoint.
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 42 | 43
days | -3.6 (0.99) | -5.1 (1.01)
Statistical Analysis 1: Comparison: Fremanezumab vs Placebo; Test type: Superiority; p = 0.1876, ANCOVA — Threshold for significance at 0.05 level; LS Mean = 1.5, 95% CI 2-sided [-0.73 to 3.67], Standard Error of Mean 1.11

2. Secondary Outcome: DB Period: Number of Participants Reaching at Least 50% Reduction From Baseline in Monthly Average Number of Headache Days of Any Severity During 12-Week Treatment With Fremanezumab
Description: Monthly averages were derived and normalized to 28 days equivalent by the following formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in the e-diary over the relevant period) * 28.
Time Frame: Baseline (Day -28 to Day-1) up to Week 12
Population: FAS included all randomized participants who received at least 1 dose of the study drug and had at least 1 post-baseline efficacy assessment on the primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 42 | 43
Participants | 5 | 4

3. Secondary Outcome: DB Period: Number of Participants Reaching at Least 50% Reduction From Baseline in the Monthly Average Number of Headache Days of at Least Moderate Severity During 12-Week Treatment With Fremanezumab
Description: A headache day was defined as a day when a participant reported a headache of at least moderate severity. Monthly averages were derived and normalized to 28 days equivalent by the following formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in the e-diary over the relevant period) * 28.
Time Frame: Baseline (Day -28 to Day-1) up to Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 42 | 43
Participants | 9 | 11

4. Secondary Outcome: DB Period: Number of Participants Reaching at Least 50% Reduction From Baseline in the Monthly Average Number of Headache Days of at Least Moderate Severity During First 4-Week (Month 1), 5- to 8-Week (Month 2), and 9- to 12-Week (Month 3)
Description: as for outcome 3
Time Frame: Baseline (Day -28 to Day-1) up to Months 1, 2, and 3
Population: FAS included all randomized participants who received at least 1 dose of the study drug and had at least 1 post-baseline efficacy assessment on the primary endpoint. Here, 'Number analyzed' signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 42 | 43
Participants
  Month 1 | 8 | 11
  Month 2: number analyzed (Participants) | 38 | 41
  Month 2 | 8 | 14
  Month 3: number analyzed (Participants) | 37 | 37
  Month 3 | 14 | 12

5. Secondary Outcome: DB Period: Change From Baseline in the Number of Headache Days of At Least Moderate Severity During the First 4-Week (Month 1), 5- to 8-Week (Month 2), and 9- to 12-Week (Month 3)
Description: A headache day was defined as a day when a participant reported a headache of at least moderate severity. Monthly averages were derived and normalized to 28 days equivalent by the following formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in the e-diary over the relevant period) * 28. The change was calculated as post-baseline value - baseline value. LS mean was calculated using ANCOVA model with the duration of post traumatic headache history (less than 12 month since the brain injury or greater or equal to 12 month since the brain injury) and treatment as fixed effects and the baseline monthly average number of headache days of at least moderate severity as a covariate. This approach was used in generating the LS mean values only and was not considered to be an additional statistical analysis, no additional statistical analyses are reported for this outcome measure.
Time Frame: Baseline (Day -28 to Day -1), up to Months 1, 2, and 3
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 42 | 43
days
  Change at Month 1 | -3.6 (0.97) | -4.0 (0.99)
  Change at Month 2: number analyzed (Participants) | 38 | 41
  Change at Month 2 | -3.7 (1.06) | -6.7 (1.06)
  Change at Month 3: number analyzed (Participants) | 37 | 37
  Change at Month 3 | -5.2 (1.20) | -7.2 (1.21)

6. Secondary Outcome: DB Period: Change From Baseline in Disability Score, as Measured by the 6-Item Headache Impact Test (HIT-6) Total Score at Week 12 After the First Dose of Fremanezumab
Description: HIT-6 is a tool used to measure the impact headaches have on a participant's normal daily life and ability to function. The HIT-6 consists of 6 items, including pain, social functioning, role functioning, vitality, cognitive functioning, and psychological distress. Each item was answered on a 5-point Likert scale (6=never, 8=rarely, 10=sometimes, 11=very often, or 13=always), which were summed to produce a total score that ranged from 36 to 78, with larger scores reflecting greater impact of headache on the daily life of the participant.
Time Frame: Baseline (Day -28 to Day -1), Week 12
Population: FAS included all randomized participants who received at least 1 dose of the study drug and had at least 1 post-baseline efficacy assessment on the primary endpoint. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 35 | 37
units on a scale | -6.9 (4.54) | -10.8 (4.65)

7. Secondary Outcome: DB Period: Number of Participants (Responder and Non-Responder) With the Patient Global Impression of Change (PGIC) Scale at Weeks 4, 8, and 12 After the First Dose of Fremanezumab
Description: The PGIC scale is a validated generic tool for the assessment of overall change in the severity of illness following treatment. Participants rated how they felt during assigned time points compared with how they felt before receiving study drug on a 7-point scale, where 1 = No change (or it got worse); 2 = Almost the same, hardly any change at all; 3 = A little better, but no noticeable change; 4 = Somewhat better, but the change has not made any real difference; 5 = Moderately better, and a slight but noticeable change; 6 = Better, and a definite improvement that has made a real and worthwhile difference; and 7 = A great deal better, and a considerable improvement that has made all the difference. Responders were those with a scale of 5 to 7 and non-responders were those with a scale of 1 to 4.
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 42 | 43
Participants
  Week 4: Responder | 12 | 11
  Week 4: Non-Responder | 24 | 26
  Week 4: Missing | 6 | 6
  Week 8: Responder | 14 | 17
  Week 8: Non-Responder | 20 | 21
  Week 8: Missing | 8 | 5
  Week 12: Responder | 11 | 16
  Week 12: Non-Responder | 20 | 16
  Week 12: Missing | 11 | 11

8. Secondary Outcome: DB Period: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were defined as AEs occurring at or after the first dose of the study drug. Serious AEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day -28 to -1) up to Week 12
Population: DB safety analysis set included all randomized participants who received at least 1 dose of study drug during the DB treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 43 | 43
Participants | 31 | 35

9. Secondary Outcome: OL Period: Number of Participants With TEAEs
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were defined as AEs occurring at or after the first dose of the study drug. Serious AEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Week 12 up to Week 24
Population: OL-ITT analysis set included only participants who received at least 1 dose of study drug during the open-label treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 9 | 7
Participants | 8 | 6

10. Secondary Outcome: DB Period: Number of Participants Who Did Not Complete the Study
Description: Number of participants who did not complete the study due to any reason and due to AEs are reported.
Time Frame: Baseline (Day -28 to Day -1) up to Week 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 43 | 43
Participants
  Discontinued study due to any reason | 15 | 17
  Discontinued study due to AEs | 1 | 1

11. Secondary Outcome: OL Period: Number of Participants Who Did Not Complete the Study
Description: Number of participants who did not complete the study due to any reason and due to AEs are reported.
Time Frame: Week 12 up to Week 24
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 9 | 7
Participants
  Discontinued study due to any reason | 1 | 1
  Discontinued study due to AEs | 0 | 0

12. Secondary Outcome: DB Period: Number of Participants Who Received Concomitant Medications
Description: Concomitant medications included: agents acting on renin-angiotensin system, analgesics, anesthetics, anti-parkinson drugs, antianemic preparations, antibacterials for systemic use, antidiarrheals, intestinal antiinflammatory/antiinfective agents, antiemetics and antinauseants, antiepileptics, antifungals for dermatologiocal use, antihistamines for systemic use, antihypertensives, antiinflammatory and antirheumatics, antineoplastic agents, antiobesity preparations, antipruritics, antithrombotics, antivirals for systemic use, beta blocking agents, calcium channel blockers, cardiac therapy, corticosteroids, cough and cold preparations, diuretics, lipid modifying agents, nasal preparations, thyroid therapy, urologicals, vaccines, psycholeptics, psycoanaleptics, ophthalmologicals, general nutrients, mineral supplements, muscle relaxants, vitamins, drugs used in diabetes, sex hormones and modulators of the genital system, immunosuppresants, drugs for acid related disorders etc.
Time Frame: Baseline (Day -28 to Day -1) up to Week 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 43 | 43
Participants | 43 | 42

13. Secondary Outcome: OL Period: Number of Participants Who Received Concomitant Medications
Description: Concomitant medications included: agents acting on renin-angiotensin system, analgesics, anti-parkinson drugs, antianemic preparations, antibacterials for systemic use, antiemetics and antinauseants, antihistamines for systemic use, antihypertensives, antiinflammatory and antirheumatics, antineoplastic agents, antithrombotics, beta blocking agents, calcium channel blockers, corticosteroids for systemic use, cough and cold preparations, diuretics, lipid modifying agents, nasal preparations, other gynecologicals, other nervous system drugs, thyroid therapy, unspecified herbal and traditional medicine, urologicals, vaccines, psycholeptics, psycoanaleptics, general nutrients, mineral supplements, muscle relaxants, vitamins, sex hormones and modulators of the genital system, drugs for acid related disorders, drugs for constipation, drugs for obstructive airways disease etc.
Time Frame: Week 12 up to Week 24
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 9 | 7
Participants | 9 | 7

14. Secondary Outcome: Number of Participants With Positive Findings on Electronic Columbia Suicide Severity Rating Scale (eC-SSRS)
Description: eC-SSRS is a questionnaire to assess suicidal ideation (severity and intensity) and behavior. Suicidal ideation: A series of 1 -5 questions (with 'yes' or 'no' response) with 5 types of ideation of increasing severity: 1. wish to be dead, 2. non-specific active suicidal thoughts, 3. active suicidal ideation with any methods (not plan) without intent to act, 4. active suicidal ideation with some intent to act, without specific plan, 5. active suicidal ideation with specific plan and intent. A positive finding was defined as a 'yes' response to question 4 or 5.
Time Frame: Baseline (Day -28 to Day -1) up to Week 24
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 43 | 43
Participants | 0 | 0

15. Secondary Outcome: Number of Participants With Treatment-Emergent Antidrug Antibodies (ADA)
Description: Number of participants with treatment-emergent antidrug antibodies reported.
Time Frame: Baseline (Day -28 to Day -1) up to Week 24
Population: ITT analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Fremanezumab | Placebo
Number analyzed (Participants) | 44 | 43
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day -28 to Day -1) up to Week 24
Description: Safety analysis set included all randomized participants who received at least 1 dose of the study drug.
Arm/Group | Fremanezumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 2/43 | 1/43
Other Adverse Events (participants affected / at risk) | 28/43 | 29/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fremanezumab (N=43) | Placebo (N=43)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fremanezumab (N=43) | Placebo (N=43)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (6) | 2 (2)
Injection site erythema (General disorders) | 11 (30) | 14 (41)
Injection site induration (General disorders) | 18 (60) | 14 (49)
Injection site pain (General disorders) | 14 (48) | 15 (47)
Injection site pruritus (General disorders) | 4 (8) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 1 (2)
Nasopharyngitis (Infections and infestations) | 2 (3) | 4 (4)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 4 (5) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (5)
International normalised ratio increased (Investigations) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 6 (7) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT03347188/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT03347188/SAP_001.pdf